CLINICAL TRIAL: NCT00182494
Title: A Five Year, Prospective, Randomized, Blinded, Controlled Trial Comparing the Efficacy of a Modified Diabetes Prevention Protocol and the Standard Comprehensive Outpatient Care in Lowering the Incidence of New Onset Diabetes Among People Treated for Schizophrenia and Are at Risk to Develop Type II Diabetes Mellitus.
Brief Title: Diabetes Prevention Program in Schizophrenia [DPPS]
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: The Lawson Foundation (Other); Ontario Mental Health Foundation (Other Government)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-2417
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-07

CONDITIONS: Diabetes Mellitus; Schizophrenia
Keywords: Schizophrenia, Diabetes, Weight gain, Antipsychotic drugs
MeSH Terms: conditions — Diabetes Mellitus; Schizophrenia; Weight Gain | interventions — Metformin

INTERVENTIONS:
Behavioral: Modified diabetes prevention protocol & Metformin

SUMMARY:
Diabetes is 2-5 times more common in schizophrenia and it is a preventable; but the current diabetes prevention guidelines are not suitable for implementation in the severely mentally ill population. The principles of diabetes prevention are essentially dietary regulation, increased physical activity and adjunctive use of oral anti-diabetic drugs (metformin). In a modified diabetes prevention protocol suitable for use in mentally ill population, we packaged the original guide lines with an adventure and recreation program based on principles of experiential learning, cognitive restructuring and behaviour modification. In this proposed study, we plan to evaluate the feasibility of adopting the new protocol, and examine its effectiveness in preventing diabetes.

DETAILED DESCRIPTION:
Rationale:

* From large international RCT studies, Type 2 Diabetes can be prevented / delayed for overweight, pre-diabetic individuals by making basic lifestyle changes (regular moderate exercise, healthy eating habits) and using metformin or other insulin resistance inhibitor.
* Individuals with schizophrenia are in particular need of preventative intervention and conventional approaches do not match their needs.
* Research has not examined how to facilitate lifestyle changes in the lives of individuals with schizophrenia.

We need to…

* Develop and evaluate innovative diabetes prevention strategies tailored to meet the needs of individuals with schizophrenia.
* Research how to make it work for pre-diabetic individuals being treated for schizophrenia.

The effectiveness of the novel intervention will be tested using a prospective, randomized, controlled clinical trial. A multi-factorial design enables a 2 x 2 analysis of the independent effects of three interventions - a tailored lifestyle modification program, metformin, and the standard conventional intervention. There is no anticipated interaction effect between metformin and lifestyle interventions. Clients currently treated for schizophrenia at a community outpatient clinic will be screened for diabetes, and those who fulfill the inclusion criteria, and give written consent, following a three week run-in period, will be randomized to one of four groups to receive either: the experimental intervention with placebo, the experimental intervention with metformin or the conventional intervention with placebo or conventional intervention with metformin.

ELIGIBILITY:
Inclusion Criteria:

1. People who are at least 18 years old, diagnosed as having schizophrenia, confirmed through a structured clinical interview (SCID-P) for DSM IV, treated with antipsychotic drugs at least for 2 years and deemed clinically stable. Clinical stability is operationally defined as absence of a relapse warranting hospitalization in the preceding six months.
2. People who are deemed as "pre-diabetics" in accordance with the diagnostic criteria established by the American Diabetic Association (ADA, 2004) as following: impaired fasting glucose (IFG) indicating fasting plasma glucose ranging between 100-125 mg/dl or 5.6 - 6.9 mmol/l.; and impaired glucose tolerance (IGT) indicating 2-h post-load glucose ranging between 140-199 mg/dl or 7.8 - 11.0 mmol/l.
3. People who have gained > 10% body weight since??? Or body mass index > 24 kg/m², except Asian decent at 22 kg/m² or greater??
4. Competent to provide informed consent to voluntarily participate in the study.

Exclusion Criteria:

1. People who meet the criteria for diabetes, (i.e., repeat fasting blood glucose (FBG) >7 mmol/l or, 2 hr. post-load glucose >11.1 mmol. as determined by a 2 hr. glucose tolerance test (GTT)).
2. People with evidence of clinically significant liver disease, renal or gastrointestinal impairments, as suggested by clinical history and liver and kidney functions tests. Any impairment deemed clinically significant would be a relative contra-indication for the use of metformin.
3. Women in the child bearing age, who are not willing to use contraceptive measures.
4. People with other comorbid disorders such as clinically significant heart or lung disease that may prevent participation in various physical activities or disorders of glucose metabolism (e.g., Cushing's Syndrome, Acromegaly, and chronic pancreatitis).
5. People with treatments that would interfere with participation or completion of the protocol (e.g., in shared care and planning to be discharged shortly from the clinic), or having a confounding effect on the measurement of the primary outcomes of the study (prescription weight loss drugs, lipid lowering agents?)
6. People with weight loss >10% in past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-02; Study Completion 2009-01

PRIMARY OUTCOMES:
1. Adherence/ability to run as designed /recruitment
2. Impact on modifiable diabetes risk factors
3. Impact on incidence of diabetes

SECONDARY OUTCOMES:
1. Adherence Rates for Diet, Exercise, Meds
2. Changes in lifestyle, Changes in eating patterns, Changes in activity patterns
3. Sustained changes in eating & activity patterns

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi P Voruganti, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada